CLINICAL TRIAL: NCT01189175
Title: Relative Bioavailability of a Single Oral Dose of BI 113823 (50 mg qd) When Administered Alone or in Combination With Multiple Oral Doses of Ketoconazole (200 mg Bid) in Healthy Male Volunteers (an Open Label, Two Periods, Fixed-sequence, Clinical Phase I Study)
Brief Title: Study in Healthy Male Subjects to Investigate Whether Ketoconazole Affects Plasma Exposure of BI 113823
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1272.5; 2010-018542-31 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

ARMS (2):
- BI 113823 (Experimental): single oral dose per subject
  Interventions: Drug: BI 113823
- BI 113823 + Ketokonazole (Experimental): after wash-out 5 days ketokonazole with BI 113823 on day 3
  Interventions: Drug: BI 113823 + Ketokonazole

INTERVENTIONS:
Drug: BI 113823 + Ketokonazole — 5 days ketokonazole with single oral dose of BI 113823 on day 3
  Arms: BI 113823 + Ketokonazole
Drug: BI 113823 — single oral dose
  Arms: BI 113823

SUMMARY:
The objective of the study is to investigate whether ketoconazole affects plasma exposure of BI 113823

ELIGIBILITY:
Inclusion criteria:

healthy male subjects

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
AUC0-∞(area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) of BI 113823 | 2 weeks
Cmax (maximum measured concentration of the analyte in plasma) of BI 113823 | 2 weeks

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | 2 weeks
Number of participants with clinically significant changes in physical examination | up to 24 days
Number of participants with clinically significant changes in vital signs | up to 24 days
Number of participants with clinically significant changes in ECG | up to 24 days
Number of participants with clinically significant changes in laboratory tests | up to 24 days
Occurrence of adverse events | up to 24 days
Assessment of tolerability by the investigator | up to 24 days
AUCt1-t2 (Area under the concentration time curve of the analyte in plasma over the time interval t1 to t2) | 2 weeks
AUC0-tmax (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to median tmax | 2 weeks
tmax (time from dosing to the maximum concentration of the analyte in plasma) | 2 weeks
λz (terminal rate constant in plasma) t1/2 (terminal half-life of the analyte in plasma | 2 weeks
t1/2 (terminal half-life of the analyte in plasma) | 2 weeks
MRTpo (mean residence time of the analyte in the body after po administration) | 2 weeks
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | 2 weeks
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | 2 weeks
Ae0-24 (amount of analyte that is eliminated in urine from the time interval 0 to 24) | visit 2, day 1 and visit 4 day 1
fe0-24 (fraction of administered drug excreted unchanged in urine from time point 0 to 24 | visit 2, day 1 and visit 4 day 1
CLR,0-24 (renal clearance of the analyte in plasma from the time point 0 until the time point 24) | visit 2, day 1 and visit 4 day 1

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1272.5.1 Boehringer Ingelheim Investigational Site, Biberach, Germany